CLINICAL TRIAL: NCT00485485
Title: Phase II Study of Imatinib Mesylate and Docetaxel in Patients With Metastatic or Recurrent Head and Neck Squamous Cell Cancer
Brief Title: Imatinib Mesylate (Gleevec) and Docetaxel in Patients With Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0362
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Head and Neck Cancer; Squamous Cell Cancer
Keywords: Head and Neck Cancer; Squamous Cell Cancer; Imatinib Mesylate; Gleevec; Imatinib; STI571; Docetaxel; Taxotere
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate + Docetaxel (Experimental): Imatinib 400 mg orally daily; Docetaxel 60 mg/m^2 by vein over 1 hour every 3 weeks
  Interventions: Drug: Imatinib Mesylate; Drug: Docetaxel

INTERVENTIONS:
Drug: Imatinib Mesylate — 400 mg by mouth daily
  Other Names: Gleevec; Imatinib; STI571
Drug: Docetaxel — 60 mg/m^2 by vein (IV) over 1 hour every 3 weeks
  Other Names: Taxotere

SUMMARY:
Primary Objective:

* To determine the efficacy of the combination of imatinib mesylate and docetaxel in recurrent or metastatic head and neck squamous cell cancer by serial measurements of tumor response (extent, frequency, duration).

Secondary Objectives:

* To assess the safety and tolerability of imatinib mesylate and docetaxel in patients with recurrent or metastatic head and neck squamous cell cancer.
* To explore the biologic effects of imatinib mesylate and docetaxel on tumor tissue by immunohistochemical analysis of microvessel density and phosphorylation of Platelet-derived growth factor receptors (PDGF-R).
* To explore the effects of imatinib mesylate and docetaxel on surrogate markers in serum.
* To assess the rate of survival.

DETAILED DESCRIPTION:
Imatinib mesylate is designed to block certain proteins important in the growth of cancer. Docetaxel is designed to target and destroy cancer cells.

If you are found to be eligible to take part in this study, you will take 4 imatinib mesylate tablets by mouth once a day with a meal and a large glass of water (about 8-10 ounces.) A treatment cycle on this study is 21 days. You should keep normal eating habits, however a low-fat breakfast is recommended (for example, a light continental breakfast of toast and juice). Foods and drinks containing caffeine or grapefruit should be avoided. You should wait at least 1 hour after taking the last tablet before going to bed. If vomiting occurs, do not take any extra study medication.

You will be given a patient diary to record when you take your medication. You should bring the diary to each clinic visit, and the study nurse will review it each time.

Docetaxel will be given through a vein in your arm on the first day of each 21-day treatment cycle for a total of 6 cycles. The infusion will take 1 hour.

You will need to take steroids (dexamethasone) before receiving docetaxel to try to prevent fluid accumulation and allergic reactions. You will take dexamethasone by mouth twice a day on the day before the docetaxel infusion, the day of the infusion, and the day after infusion. You will receive an extra dose of dexamethasone (either through a needle in a vein or by mouth) on the day of infusion of the chemotherapy either through a needle in a vein or by mouth.

Every 3 weeks while on this study, you will have a physical exam, including measurement of your vital signs and weight, and a performance status evaluation. During the first 4 weeks, blood (about 3 teaspoons each time) will be drawn once a week for routine tests. After that, blood (about 3 teaspoons each time) will be drawn once at Week 5, once at Week 7, and then every 3 weeks after that. In addition, your tumor will be measured by a computed tomography (CT) or magnetic resonance imaging (MRI) scan every 6 weeks (at Weeks 7, 13, and 19).

If you develop any intolerable symptoms or certain changes in your blood tests, your treatment may be delayed and/or the dose may be decreased until the symptoms are gone. It may even be necessary to stop your treatment. You will be informed of any changes in your dosing schedule or in the doses of your medication after your doctor evaluates you in the clinic.

You may receive up to 6 cycles of the study treatment. Your continued participation in this study depends on how the cancer responds to the study drugs. Your doctor may decide to take you off this study if you experience intolerable side effects or the medical condition gets worse.

After you have completed all of your treatment, you will have an end-of-study visit. At this visit you will have a physical exam, including measurement of your vital signs and weight. You will have a performance status evaluation. You will have blood (about 3-4 teaspoons) drawn for routine tests. Your tumor will be measured by a CT or MRI scan.

This is an investigational study. Imatinib mesylate is FDA approved and docetaxel are FDA approved for other types of cancer however their use together in this study is investigational. Dexamethasone is required to be given with docetaxel. All three drugs are commercially available. Up to 58 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A written, voluntary informed consent form must be completed prior to beginning any study procedure.
2. Patients >/= 18 years of age.
3. Histologically documented diagnosis of head and neck squamous cell cancer
4. At least one measurable site of disease and can be assessed by Response Evaluation Criteria In Solid Tumors (RECIST).
5. Performance status 0-2 (Eastern Cooperative Oncology Group, ECOG)
6. Patients must have adequate hepatic, renal, and bone marrow function, defined as the following: (1) total bilirubin < 1.5 * Upper Limits of Normal (ULN); (2) aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) < 2.5 * ULN; (3) creatinine < 1.5 * ULN; (4) ANC > 1.5 * 10^9/L; (5) platelets > 100 * 10^9/L.
7. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control (i.e. condoms, diaphragm) throughout the study and for up to 3 months following discontinuation of study drug.
8. Patients who have not been treated for recurrent or metastatic head and neck squamous cell carcinomas (HNSCC) (i.e. Patients who have been treated with chemotherapy for induction/adjuvant or concurrent therapy with radiation in the setting of definitive treatment but have now developed recurrent or metastatic disease are eligible).

Exclusion Criteria:

1. Prior exposure to docetaxel or imatinib mesylate.
2. Patient has received any other investigational agents within 30 days of first day of study drug dosing.
3. Patients with myocardial infarction within the past 6 months or New York Heart Association class 3 or 4 congestive heart failure.
4. Female patients who are pregnant or breast-feeding.
5. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection (i.e. septic).
6. Patient has unstable brain metastasis. Unstable brain metastasis is defined as patients on steroid medication to control symptoms or patient with motor neurologic compromise due to brain metastasis. Patients with treated brain metastasis are eligible if they are > 6 weeks out from therapy and off all steroid medication.
7. Patient has known chronic liver disease (i.e., chronic active hepatitis or cirrhosis).
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection. HIV patients are at much greater risk of infection when receiving highly myelosuppressive agents (docetaxel and imatinib) and for safety reasons are not eligible for this trial.
9. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
10. Patient previously received radiotherapy to >/= 25 % of the bone marrow
11. Patient had a major surgery within 2 weeks prior to study entry.
12. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
13. Patients must agree not to use herbal remedies or other over-the-counter biologics (i.e. shark cartilage)
14. History of hypersensitivity to docetaxel or other taxane therapy.
15. History of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
16. Patients taking therapeutic levels of warfarin. However, patients receiving 1 mg daily for catheter related anticoagulation are eligible for the study.
17. Prior pericardial effusion requiring intervention such as pericardiocentesis or pericardial window within 2 months of study entry.
18. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
19. Patients with a history of Regional Ileitis, Colitis, or Crohn's disease, or any other relevant medical history related to the integrity of the bowel wall as there may be an increased risk of bowel perforation with the combination of Docetaxel and Imatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S. Tsao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall Study Recruitment: 1/18/2007 - 3/18/2008. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Patient has received any other investigational agents within 30 days of first day of study drug dosing; Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
Period: Overall Study
Arm/Group | Imatinib Mesylate + Docetaxel
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate + Docetaxel
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Participant Response Rate
Description: Response rate to regimen defined as the number of complete or partial response divided by the total number of participants treated. Tumor response defined by Response Evaluation Criteria In Solid Tumors (RECIST). All complete and partial responses confirmed by a second assessment six weeks later.
Time Frame: At 6 weeks reconfirmed 6 weeks later
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate + Docetaxel
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Study Period of 3 years, one month (1/18/2007 - 2/24/2010)
Arm/Group | Imatinib Mesylate + Docetaxel
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate + Docetaxel (N=7)
Neutropenic Fever (Infections and infestations) | 1 (2)
PEG SITE INFECTION G3 (Infections and infestations) | 1 (1)
ANEMIA G3 (Blood and lymphatic system disorders) | 1 (3)
Swelling G3 (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Renal and urinary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Thrombocytopenia (Grade 3) (Blood and lymphatic system disorders) | 1 (1)
Mucositis G3 (Gastrointestinal disorders) | 1 (3)
Dysphagia G3 (Gastrointestinal disorders) | 1 (3)
Palpitations (Cardiac disorders) | 1 (1)
Cardiovascular Pain (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate + Docetaxel (N=7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Edema: Head and Neck (Blood and lymphatic system disorders) | 2 (2)
Bilirubin (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophils (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was closed to enrollment early due to low enrollment. Study enrolled 7 participants over approximately 2 years with a planned enrollment of up to 58.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No